CLINICAL TRIAL: NCT00986427
Title: Restasis® Ophthalmic Emulsion for the Treatment of Brittle Nails
Brief Title: Restasis for Treatment of Brittle Nails
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Julian M. Mackay-Wiggan (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Julian M. Mackay-Wiggan, Assistant Clinical Professor of Dermatology, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAD9927; Res-01-2009 (Other: Protocol number)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-07

CONDITIONS: Brittle Nails
MeSH Terms: conditions — Twenty-Nail Dystrophy | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects will apply Restasis® to the target nails for 24 weeks. Additionally, there is a 12 week follow up period post the treatment period.
  Interventions: Drug: Restasis (cyclosporine ophthalmic emulsion) 0.05%
- 2 (Placebo Comparator): Subjects will apply Refresh® Dry Eye therapy to the target nails for 24 weeks. Additionally, there is a 12 week follow up period post the treatment period.
  Interventions: Drug: Refresh® Dry Eye therapy

INTERVENTIONS:
Drug: Restasis (cyclosporine ophthalmic emulsion) 0.05% — cyclosporine ophthalmic emulsion 0.05%
  Other Names: Restasis®
  Arms: 1
Drug: Refresh® Dry Eye therapy — Emulsion contains glycerin 1% and polysorbate 80
  Other Names: Refresh®
  Arms: 2

SUMMARY:
This purpose of this study is to assess the safety and effectiveness of Restasis® ophthalmic emulsion versus emulsion alone( Refresh Dry Eye therapy) both for the treatment of brittle nails and for the enhancement of normal nail growth and texture. The investigators think that daily application of Restasis® to nails and nail beds in patients with brittle nails will enhance nail growth and improve nail texture in both affected and unaffected nails.

DETAILED DESCRIPTION:
This is a single center, investigator-blinded (investigator masked), head to head comparison of Restasis® and its vehicle, Refresh® Dry Eye Therapy in 24 patients. Three target fingernails will be identified in each subject. Two of the target nails will be the two nails that have the most severe signs of brittle nail syndrome. The third target nail will be a normal nail or, in the absence of a normal nail, the patient's second-healthiest appearing nail. The patients most normal-appearing nail will be untreated so that growth in the treated nails can be compared to growth in an untreated normal nail, this will be the fourth target nail. Study medication will be applied to target nails (the subjects may also apply to all nails if they wish, except one nail which will be untreated in order to determine the subject's baseline rate of fingernail growth) for 24 weeks. The target nails will be assessed at each visit, every four weeks. There will be a 12-week follow up period after treatment is completed.

This 36 week study will be conducted at one center. Adult male and female patients meeting the inclusion and exclusion criteria will be screened for eligibility. The principal investigator or his/her designee will obtain informed consent from all patients before any protocol specific procedures are performed.

ELIGIBILITY:
Inclusion Criteria:

* must have IRB approved written informed consent prior to participating in any study related procedures
* Must be a male or female patient 18 to 75 years of age
* must have a diagnosis of brittle or meet the criteria for a diagnosis of brittle nails at the screening visit based on at least two of the following signs and symptoms of brittle nails in each of the selected nail plates or severe signs (one or more) on each target nail
* trachyonychia (surface roughness)
* lamellar onychoschizia (horizontal layering/peeling
* longitudinal cracking or splitting of the distal edge (raggedness)
* must have two fingernails with brittle nail signs and symptoms identified at baseline
* must have two normal or near-normal nails on the same hand
* female patients of childbearing potential (not surgically sterile or at least 2 years postmenopausal) must have a negative pregnancy at baseline/day 1 and may not be lactating
* sexually active female subjects who are not surgically sterile or 2 years post menopausal must agree to use contraception/birth control measure while on study (e.g., oral contraceptive, diaphragms with spermicide, condoms with spermicide, intrauterine devices, Norplant System, Depo-Provera, tubal ligation). Monthly urine pregnancy tests will be administered to women of childbearing potential
* must agree to self administer topical study medication, and must agree to complete all study procedures
* must be judged to be in good health by medical history and physical examination
* must be able to adhere to the study visit schedule and other protocol requirements, including avoiding the use of nail polish, adhesive nails, and manicures for the duration of the study

Exclusion Criteria:

* have a history of surgery of the affected fingernails
* are chronic nail biters
* are pregnant, nursing, or planning pregnancy prior to study enrollment
* have a disturbance of the shape of the affected fingernails (e.g., due to malformation of the underlying bone) that would interfere with the investigator's ability to evaluate photographs or nail changes
* have onycholysis (lifting of the nail plate off the nail bed) of the affected fingernails
* have signs of a fungal or bacterial infection of the affected fingernails
* have a history of psoriasis or lichen planus involving any nail, or active contact dermatitis involving the affected fingernails
* have used any topical cosmetics or medicated products on the affected nails within 2 weeks of baseline visit
* have received oral antifungal treatment within 3 months of baseline visit
* have a known or suspected history of a genetic condition affecting the nails (e.g., Darier's disease, nail-patella syndrome, tuberous sclerosis)
* have used any investigational drug within the previous 1 month or 5 half-lives of the investigational agent, whichever is longer, or 3 months for any biologic of unknown half-life
* are known or suspected to have had a substance abuse (drug or alcohol) problem within the previous 3 years
* is unlikely to comply with the study protocol and prescribed treatment or is unsuitable for any other reason in the opinion of the investigator
* chronic liver, heart, kidney, or (untreated) thyroid disease
* have current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease
* currently have any known malignancy or have a history of malignancy other than non-melanoma skin cancer
* have signs of bacterial, fungal or viral skin lesions that may interfere with evaluation of the target nails
* known sensitivity to any active or inactive ingredient in Restasis(R) or Refresh(R) Dry Eye Therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Mackay Wiggan, MD, MS, Principal Investigator — Columbia University Medical Center Department of Dermatolgoy
Locations (1):
- Columbia University Medical Center Department of Dermatology, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 patients recruited.
Groups:
- Restasis® Arm: Subjects will apply Restasis® to the target nails for 24 weeks. Additionally, there is a 12 week follow up period post the treatment period.
- Refresh® Arm: Subjects will apply Refresh® Dry Eye therapy to the target nails for 24 weeks. Additionally, there is a 12 week follow up period post the treatment period.
Period: Overall Study
Arm/Group | Restasis® Arm | Refresh® Arm
Started | 12 | 12
Completed | 8 | 12
Not Completed | 4 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restasis® Arm | Refresh® Arm | Total
Number analyzed (Participants) | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (49.40) | 59.6 (12.69) | 59.7 (13.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Physician's Global Assessment (PGA) of Target Fingernails #1 and #2
Description: Change from baseline in the Physician's Global Assessment (PGA) of target fingernails #1 and #2 as measured at week 24.
  The PGA is a static evaluation/measure of the severity of brittle nails signs in target fingernails #1 and #2 (the 2 nails with the most severe signs of brittleness). Evaluated sings were the degree of lamellar onychoschizia, ridging, longtitudinal splitting, fragility/breakage and thickness. The PGA was scored on a 6 point scale from 0 to 5, in which 0 = none, 1 = mild, 2 = mild to moderate, 3 = moderate, 4 = moderate to severe, 5 = severe. A negative number change from baseline (decrease in grade score) indicates improvement and a positive change (increase in grade score) indicates worsening.
Time Frame: Baseline, week 24
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Restasis® Arm | Refresh® Arm
Number analyzed (Participants) | 12 | 12
scores on a scale | -1.4 (0.90) | -1.4 (0.67)

2. Secondary Outcome: Change From Baseline in Quality of Life (QOL) Related to Nail Disease
Description: Change from baseline in quality of life as measured at week 24 by the subject satisfaction Questionnaire question: "Overall, how satisfied are you with your nails?" Responses ranged from 1 (very satisfied) to 5 (very unsatisfied). A negative number changed from baseline (decrease in grade score) indicates improvement and a positive change (increase in grade score) indicates worsening.
Time Frame: Baseline, week 24
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Restasis® Arm | Refresh® Arm
Number analyzed (Participants) | 12 | 12
scores on a scale | -1.6 (1.19) | -0.9 (1.97)

3. Secondary Outcome: Growth of the Treated and Untreated Nail in the Previous 4 Weeks
Description: Growth of the treated and untreated nail the previous 4 weeks. Nail growth was measured in millimeters.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Groups:
- Restasis® Arm Treated Nail: Restasis® Treated Nail
- Restasis® Arm Untreated Nail: Restasis® Untreated Nail
- Refresh® Dry Eye Treated Nail: Refresh® Dry Eye Therapy Treated Nail
- Refresh® Dry Eye Untreated Nail: Refresh® Dry Eye Therapy Untreated Nail
Arm/Group | Restasis® Arm Treated Nail | Restasis® Arm Untreated Nail | Refresh® Dry Eye Treated Nail | Refresh® Dry Eye Untreated Nail
Number analyzed (Participants) | 12 | 12 | 12 | 12
Millimeters (mm) | 3.1 (1.36) | 2.9 (1.83) | 2.9 (1.15) | 2.7 (0.62)

4. Secondary Outcome: Number of Subjects Achieving Improvement in the Physician's Global Improvement Assessment (PGIA)
Description: Number of subjects achieving improvement in the PGIA. The investigator assessed the two target fingernails with a rating of Excellent, Good, Fair, No Improvement or Worse based on the comparison between the nails at the current visit and high-resolution photographs of the nails taken at baseline. An improvement was a score of Excellent/Good/Fair vs. No Improvement/Worse.
Time Frame: Week 24
Measure: Number; unit: participants
Arm/Group | Restasis® Arm | Refresh® Arm
Number analyzed (Participants) | 12 | 12
participants | 10 | 9

ADVERSE EVENTS:
Arm/Group | Restasis® Arm | Refresh® Arm
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 9/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restasis® Arm (N=12) | Refresh® Arm (N=12)
Hematemasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Restasis® Arm (N=12) | Refresh® Arm (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Dry eye symptom (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Flu signs and symptoms (General disorders) | 1 (1) | 0 (0)
Hematemasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inflammation of right shoulder (from a fall) (General disorders) | 1 (1) | 0 (0)
Pain from car accident (General disorders) | 1 (1) | 0 (0)
Pain in both notched nails (General disorders) | 1 (1) | 0 (0)
Pain in right thumb nail (General disorders) | 1 (1) | 0 (0)
Tooth abscess - pain (General disorders) | 1 (1) | 0 (0)
Infection in the right gum (Infections and infestations) | 0 (0) | 1 (1)
Nail infection - right middle finger (cat bite) (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Stomach virus (Infections and infestations) | 0 (0) | 2 (2)
Strep throat (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Back Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small Sample Size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No